CLINICAL TRIAL: NCT00437866
Title: Hepcidin in the Pathogenesis of Anemia in Patients With Chronic Heart Failure
Brief Title: Hepcidin in Anemic Chronic Heart Failure (CHF) Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Martin Huelsmann, PI, Doctor, Medical University of Vienna
Other Study IDs: Version 1.0, 25.11.2006
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Anemia; Chronic Heart Failure
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background: Anemia in chronic heart failure (CHF) is directly linked to increased mortality and reduced exercise capacity. The pathomechanism for the development of anemia in CHF is not well understood. Impairment of iron homeostasis is discussed to be one of the major triggers in anemia of chronic disease. Hepcidin was recently described as the central regulator of iron homeostasis.

Main hypothesis: Plasma hepcidin levels are altered in anemic CHF patients compared to non anemic controls and might be a main contributing factor of anemia in CHF.

Iron regulator-hypothesis High levels of cytokines in CHF patients cause up-regulation of hepcidin, which in turn leads to low iron uptake causing anemia. In this case venous hepcidin and hemoglobin concentrations should both correlate with cytokine levels.

Erythropoietin regulator-hypothesis Dysregulation of the erythropoietin system results in anemia, which represses hepcidin. This leads to a negative correlation between hemoglobin and hepcidin in plasma.

Methods: 100 consecutive patients diagnosed with systolic CHF will be prospectively included in the study. Iron status will be assessed and hepcidin, erythropoietin as well as interleukin-1, interleukin-6 and soluble TNF alpha receptor levels will be measured by ELISA.

Patients will be followed up for one year and mortality, rehospitalization and worsening of CHF will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Systolic left ventricular dysfunction (LVEF<45%)
2. Signed informed consent

Exclusion Criteria:

1. Women of child bearing potential
2. Pregnancy
3. Non cardiac illness limiting life expectancy to <1 year
4. Renal disease of non-cardiac reason
5. Malignancy
6. Chronic inflammatory disease
7. Acute infection
8. Erythropoietin therapy or iron substitution within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart failure outpatients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Hemodilution

CONTACTS AND LOCATIONS:
Overall Officials: Martin Huelsmann, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna-Austria, Austria

REFERENCES:
- [Result] Adlbrecht C, Kommata S, Hulsmann M, Szekeres T, Bieglmayer C, Strunk G, Karanikas G, Berger R, Mortl D, Kletter K, Maurer G, Lang IM, Pacher R. Chronic heart failure leads to an expanded plasma volume and pseudoanaemia, but does not lead to a reduction in the body's red cell volume. Eur Heart J. 2008 Oct;29(19):2343-50. doi: 10.1093/eurheartj/ehn359. Epub 2008 Aug 12. PMID 18701467